CLINICAL TRIAL: NCT00904917
Title: Children of Depressed Mothers: Culture & Prevention
Brief Title: Preventing Depression in the Children of Depressed African American Mothers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rhonda Boyd, Associate Professor, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2004-10-4041; K01MH068619 (NIH); DSIR 8K-RTCT (Other: NIMH DSIR); IRB NO: 2004-10-4041 (Other: IRB No.)
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Depression
Keywords: African American Mothers; Children; African American Families; Parental Depression; Preventive Intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adapted PIP (Experimental): Participants (both mother and children) participated in an adapted cognitive family prevention program for the families of children with a depressed African American mother.
  The intervention was the Prevention Intervention Project.
  Interventions: Behavioral: Prevention Intervention Project
- Lecture (Active Comparator): Mothers received psychoeducation about depression.
  The intervention was psychoeducation.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Prevention Intervention Project — Eight 1-hour sessions focused on psychoeducation, coping with stress, and cognitive-behavioral strategies. The sessions were tailored as required to meet the clinical and cultural needs of each family; other family members, such as fathers, spouses, and grandparents, were invited to participate in the intervention.
  Arms: Adapted PIP
Behavioral: Psychoeducation — Two 1-hour sessions focusing on psychoeducation about depression and its impact on children and the family.
  Arms: Lecture

SUMMARY:
The purpose of the study is to adapt and test the Preventive Intervention Project for urban African American mothers with depression and their children.

DETAILED DESCRIPTION:
Abstract

Background: There is limited representation of ethnic minorities in preventive interventions for the generational impact of maternal depression.

Methods: The Preventive Intervention Project (PIP) was adapted to be culturally and contextually relevant for urban African American mothers with depression and their children. A pilot clinical trial (PIP vs. lecture) was conducted.

ELIGIBILITY:
Mothers:

Inclusion Criteria:

* African American
* Primary current or past-year diagnostic and statistical manual (DSM-IV) diagnosis of Major Depressive Disorder, Dysthymic Disorder, or Depressive Disorder not otherwise specified
* Parent or guardian and primary caregiver of a child 8 to 14 years old
* Resided at least part time for the past year with the targeted child
* May be receiving psychopharmacological treatment, psychosocial services, or both

Exclusion Criteria:

* Current or lifetime history of schizophrenia
* Current or lifetime history of bipolar disorder
* Current or past-year diagnosis of alcohol or drug dependency
* Serious medical disorder, neurological disorder, condition, or chronic pain that prevents participation
* Documented mental retardation
* Current suicide risk sufficient to preclude outpatient treatment

Children:

Inclusion Criteria:

* Have an African American mother with a depressive disorder
* 8 to 14 years old
* Reside at least part time with mother

Exclusion Criteria:

* Currently in treatment for depression or an anxiety disorder
* Presence of a medical or psychiatric condition contraindicating study intervention, such as mental retardation, suicidality, or pervasive developmental disorder

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda C. Boyd, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The majority of the mothers were recruited through newspaper ads while remaining participants were recruited from word of mouth, research studies, mental health clinics and other sources.
Pre-assignment Details: Eighteen mothers completed the Structured Clinical Interview (SCID), with 16 being eligible to participate in the study, and 1 mother did not complete the baseline interview. Fifteen mothers (with 19 children) were randomized.
Groups:
- Adapted PIP (Mothers): Mothers participated in an adapted PIP for the families of children with a depressed African American mother.
  Prevention Intervention Project : Eight 1-hour sessions, tailored as required to meet the clinical and cultural needs of each family. Intervention focuses on education, coping with stress, and cognitive-behavioral strategies.
- Adapted PIP (Children): Children of the mother-child dyad in the adapted PIP intervention for families of children with a depressed African American Mother.
  Intervention Project: Eight 1 hour sessions, tailored as required to meet the clinical and cultural needs of each family. Intervention focuses on education, coping with stress, and cognitive-behavioral strategies
- Lecture (Mothers): Mothers who received education about depression.
  Psychoeducation : Two 1-hour sessions focusing on psychoeducation about depression and its impact on children and the family.
- Lecture (Children): Children of mothers who received education about depression.
  Psychoeducation : Two 1-hour sessions focusing on psychoeducation about depression and its impact on children and the family.
Period: Overall Study
Arm/Group | Adapted PIP (Mothers) | Adapted PIP (Children) | Lecture (Mothers) | Lecture (Children)
Started | 7 | 11 | 8 | 8
Completed | 5 | 9 | 6 | 6
Not Completed | 2 | 2 | 2 | 2
Not completed — Lost to Follow-up | 2 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The participant flow module is based on the number of mother-child dyads that completed the baseline assessment(s), while the overall number of participants is based on the number of mothers and children in the intervention and control groups.
Groups:
- Adapted PIP (Mothers): Mothers of the mother-child dyad in the adapted PIP intervention.
- Adapted PIP (Children): Children of the mother-child dyad in the adapted PIP intervention.
- Lecture (Mothers): Mothers of the mother-child dyad in the lecture control group.
- Lecture (Children): Children of the mother-child dyad in the lecture control group.
- Total: Total of all reporting groups
Arm/Group | Adapted PIP (Mothers) | Adapted PIP (Children) | Lecture (Mothers) | Lecture (Children) | Total
Number analyzed (Participants) | 7 | 11 | 8 | 8 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 11 | 0 | 8 | 19
  Between 18 and 65 years | 7 | 0 | 8 | 0 | 15
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 8 | 8 | 29
  Male | 0 | 5 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 7 | 11 | 8 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Children Depression Inventory (CDI)
Description: Children Depression Inventory (CDI; Kovacs, 1992) is a widely-used self-report scale of depressive symptoms suitable for use by youth ranging from 7 to 17 years. The CDI is a 27-item scale that is self-rated and symptom-oriented. The 27 items on the assessment are grouped into five major factor areas. The item score are rated 0-2 with a total scores summed and converted to T scores. The total T score ranges from 33 to 100 with high scores indicating higher levels of depressive symptoms.
Time Frame: Measured at baseline and at post-treatment (8 weeks after baseline)
Population: These scores are based on the CDI which was administered solely to the children of the dyadic mother-child intervention and control groups. Post-intervention scores based on 9 children in Adapted PIP (2 lost to follow-up) and 6 children in Lecture group (2 lost to follow-up).
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Adapted PIP | Lecture
Number analyzed (Participants) | 11 | 8
T scores
  Baseline scores | 47.64 (8.36) | 47.00 (8.55)
  Post-intervention scores (8 weeks from baseline) | 42.11 (2.98) | 43.83 (5.27)
Statistical Analysis 1: Comparison: Adapted PIP vs Lecture; Test type: Superiority or Other; p = .015, t-test, 2 sided

2. Primary Outcome: Multidimensional Anxiety Scale for Children (MASC)
Description: Multidimensional Anxiety Scale for Children (MASC; March et al., 1997) is a self-report instrument that measures a broad range of anxiety symptoms in youth. The MASC consists of 39 items using a 4-point Likert scale that are distributed across four major factors, three of which can be parsed into two subfactors each. Main and subfactors include (1) physical symptoms (tense/restless and somatic/autonomic), (2) social anxiety (humiliation/rejection and public performance fears), (3) harm avoidance (perfectionism and anxious coping), and (4) separation anxiety. Scores are summed and converted to T-scores. The total T score ranges from 25 to 90 with higher scores representing greater levels of anxiety.
Time Frame: Measured at baseline and post-treatment (8 weeks after baseline)
Population: These scores are based on the MASC which was administered solely to the children of the dyadic mother-child intervention and control groups. Post-intervention scores based on 9 children in Adapted PIP (2 lost to follow-up) and 6 children in Lecture group (2 lost to follow-up).
Measure: Mean (Standard Deviation); unit: T scores
Arm/Group | Adapted PIP | Lecture
Number analyzed (Participants) | 11 | 8
T scores
  Baseline scores | 50.64 (8.43) | 52.50 (10.07)
  Post-intervention scores (8 weeks from baseline) | 43.67 (15.12) | 57.67 (32.36)

3. Secondary Outcome: Understanding Mood Disorders Questionnaire (UMDQ)
Description: Understanding Mood Disorders Questionnaire (UMDQ; Gavazzi, Fristad, & Law, 1997) measures attributions and knowledge of symptoms, course, and treatment of mood disorders and a symptom checklist. It has 39 items and two subscales. A range of total score is 0 to 59. The first 20 questions are true/false questions and correct responses are scored 2 points each. Nineteen questions are a checklist of symptoms and correct identification of those depression and manic symptoms are scored 1 point each. All items are summed for a total score. Higher scores indicate greater knowledge of mood disorders. Both maternal and child reporters completed this measure.
Time Frame: Measured at baseline and post-treatment (8 weeks after baseline)
Population: These scores are based on the UMDQ, which was administered to both the mothers and their children of the dyadic mother-child intervention and control groups. Post-intervention scores based on 5 mothers and 9 children in Adapted PIP (4 participants lost to follow-up) and 6 mothers and 6 children in Lecture group (4 participants lost to follow-up).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adapted PIP (Mother); Adapted PIP (Child): Participants (both mother and children) participated in an adapted cognitive family prevention program for the families of children with a depressed African American mother.
  The intervention was the Prevention Intervention Project.
- Lecture (Mother): Mothers received psychoeducation about depression.
- Lecture (Child): Mothers received psychoeducation about depression. The intervention was psychoeducation.
Arm/Group | Adapted PIP (Mother) | Adapted PIP (Child) | Lecture (Mother) | Lecture (Child)
Number analyzed (Participants) | 7 | 10 | 8 | 8
units on a scale
  Baseline scores | 23.86 (3.93) | 14.70 (5.72) | 24.25 (3.41) | 13.13 (5.57)
  Post-intervention scores (8 weeks from baseline) | 22.80 (2.59) | 14.67 (5.45) | 25.00 (2.10) | 14.33 (4.18)
Statistical Analysis 1: Comparison: Adapted PIP (Child) vs Lecture (Child); Test type: Superiority or Other; p = .037, Regression, Linear

4. Secondary Outcome: Child's Report on Parental Behavior Inventory (CRPBI)
Description: Child's Report on Parental Behavior Inventory (CRPBI; Schludermann & Schludermann, 1970) assesses children's and parents' perceptions of parental acceptance, permitting psychological autonomy, and level of parental control. The 10-item acceptance scale which assesses parental warmth was administered. The acceptable scale has items scored from 1 to 3 (not like me, somewhat like me, a lot like me). Items are summed with a total range is 10 to 30. Higher scores represents greater warmth exhibited by mother to child. Separate forms are available for both child and parent report.
Time Frame: Measured at baseline and post-treatment (8 weeks after baseline)
Population: These scores are based on the CRPBI, which was administered to both the mothers and their children of the dyadic mother-child intervention and control groups. Post-intervention scores based on 5 mothers and 9 children in Adapted PIP (4 participants lost to follow-up) and 6 mothers and 6 children in Lecture group (4 participants lost to follow-up).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lecture (Mother); Lecture (Child): Mothers received psychoeducation about depression. The intervention was psychoeducation.
Arm/Group | Adapted PIP (Mother) | Adapted PIP (Child) | Lecture (Mother) | Lecture (Child)
Number analyzed (Participants) | 7 | 11 | 8 | 8
units on a scale
  Baseline scores | 25.57 (3.21) | 24.55 (4.63) | 24.88 (4.09) | 27.13 (2.17)
  Post-intervention scores (8 weeks from baseline) | 26.40 (3.36) | 24.67 (3.46) | 25.33 (4.68) | 25.00 (4.98)

ADVERSE EVENTS:
Time Frame: Adverse event was collected for 1 year.
Groups:
- Adapted PIP: Participants (both mother and children) participated in an adapted cognitive family prevention program for the families of children with a depressed African American mother. The intervention was the Preventive Intervention Project.
- Lecture: Mothers received psychoeducation about depression.
Arm/Group | Adapted PIP | Lecture
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

LIMITATIONS AND CAVEATS:
Small sample size; Inadequate power to detect changes between groups; No-intervention comparison group; Differential attrition in the two groups favoring the comparison group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No